CLINICAL TRIAL: NCT03706066
Title: An Observational, Prospective, Post-Marketing Clinical Study of the ACRYSOF® IQ PanOptix Multifocal IOL in an Indian Population
Brief Title: India PanOptix Post Marketing Study
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ILD432-P001; CTRI/2018/11/016467 (Other: CTRI)
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PanOptix: Cataract surgery with implantation of Acrysof IQ PanOptix IOL
  Interventions: Device: Acrysof IQ PanOptix IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: Acrysof IQ PanOptix IOL — Single-piece, ultraviolet and blue-light filtering, foldable, multifocal intraocular lens (IOL) inserted into the capsular bag during cataract surgery
  Other Names: Model TFNT00
Procedure: Cataract surgery — Per investigator's standard of care

SUMMARY:
The purpose of this Post Marketing Study is to study the safety and effectiveness of the ACRYSOF IQ PanOptix intraocular lens (IOL) in an Indian population.

DETAILED DESCRIPTION:
The study population will consist of adult Indian males and females, at least 18 years of age or older at the time of screening, with no ocular pathology that could confound study outcomes, who are advised bilateral cataract extraction and who desire an IOL that provides the potential for correction of near, intermediate, and distance vision. Both eyes will be implanted. The second eye surgery will take place 15-30 days after the first eye surgery. Subjects will be followed for approximately 3 months after the second eye surgery. Total individual subject participation will be approximately 4 months. This study will be conducted in India.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures;
* Advised cataract extraction in both eyes and agreed for bilateral implantation of ACRYSOF IQ PanOptix lens;
* Preoperative regular keratometric astigmatism of ≤1.0 D in both eyes.

Exclusion Criteria:

* Pregnant or lactating, current or planned, during the course of the study;
* Retinal abnormalities (Macular Degeneration, dystrophy, edema , traction or other pathologies affecting vision);
* Clinically significant corneal abnormalities;
* History of retinal conditions;
* Previous refractive surgery, including LASIK;
* Glaucoma;
* Any condition that may not be appropriate to this study, as per the Investigator's expert medical opinion.

Other protocol-specified inclusion and/or exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll males and females who are at least 18 years of age or older at the time of screening, have no ocular pathology that could confound study outcomes, have been advised bilateral cataract extraction, and desire an intraocular lens (IOL) that provides the potential for correction of near, intermediate, and distance vision.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Best corrected binocular visual acuity at distance (4 m) at 3 months post bilateral implantation | Month 3 (following second eye surgery)
  Visual acuity will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) charts and reported in logarithm minimum angle of resolution (logMAR).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Alcon Laboratories (India) PVT.LTD
Locations (5):
- India (5):
  - Alcon Investigative Site, Ahmedabad, Gujarat
  - Alcon Investigative Site, Chennai, Tamil Nadu
  - Alcon Investigative Site, Coimbatore, Tamil Nadu
  - Alcon Investigative Site, Bangalore
  - Alcon Investigative Site, Hyderabad

IPD SHARING:
Plan to Share IPD: No